CLINICAL TRIAL: NCT02590432
Title: An Open-label, Long-term Study to Assess the Immunogenicity of Linaclotide Administered Orally to Adult Patients With Irritable Bowel Syndrome With Constipation or Chronic Idiopathic Constipation.
Brief Title: An Open-Label, Long-term Study to Assess the Immunogenicity of LINZESS® (Linaclotide) Administered Orally to Adult Participants With Irritable Bowel Syndrome With Constipation or Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIN-MD-10
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Irritable Bowel Syndrome With Constipation; Chronic Idiopathic Constipation
Keywords: Immunogenicity; Irritable Bowel Syndrome with Constipation; Chronic Idiopathic Constipation; Linaclotide; Linzess
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- LINZESS® 145 μg (CIC, Open Label) (Experimental): LINZESS® (linaclotide) 145 μg capsules, orally, once daily for up to 52 weeks for participants with CIC. If an intolerable AE occurred participants could be randomized to the Double-blind Treatment Period.
  Interventions: Drug: Linaclotide
- LINZESS® 290 μg (IBS-C, Open Label) (Experimental): LINZESS® 290 μg capsules, orally, once daily for up to 52 weeks for participants with IBS-C. If an intolerable AE occurred participants could be randomized to the Double-blind Treatment Period.
  Interventions: Drug: Linaclotide
- LINZESS® 290 μg (IBS-C, Double Blind) (Experimental): Following participation in the Open Label Treatment Period, LINZESS® 290 μg capsules, orally, once daily from double-blind randomization up to Week 52 for participants with IBS-C. If an intolerable AE occurred, dose was reduced to Open Label 72 μg, if applicable.
  Interventions: Drug: Linaclotide
- LINZESS® 145 μg (IBS-C, Double Blind) (Experimental): Following participation in the Open Label Treatment Period, LINZESS® 145 μg capsules, orally, once daily from double-blind randomization up to Week 52 for participants with IBS-C. If an intolerable AE occurred, dose was reduced to Open Label 72 μg, if applicable.
  Interventions: Drug: Linaclotide
- LINZESS® 72 μg (IBS-C, Double Blind) (Experimental): Following participation in the Open Label Treatment Period, LINZESS® 72 μg capsules, orally, once daily from double-blind randomization up to Week 52 for participants with IBS-C. If an intolerable AE occurred, dose was maintained at Open Label 72 μg, if applicable.
  Interventions: Drug: Linaclotide
- LINZESS® 145 μg (CIC, Double Blind) (Experimental): Following participation in the Open Label Treatment Period, LINZESS® 145 μg capsules, orally, once daily from double-blind randomization up to Week 52 for participants with CIC. If an intolerable AE occurred, dose was reduced to 72 μg, if applicable.
  Interventions: Drug: Linaclotide
- LINZESS® 72 μg (CIC, Double Blind) (Experimental): Following participation in the Open Label Treatment Period, LINZESS® 72 μg capsules, orally, once daily from double-blind randomization up to Week 52 for participants with CIC. If an intolerable AE occurred, dose was maintained at Open Label 72 μg, if applicable.
  Interventions: Drug: Linaclotide
- LINZESS® 72 μg (CIC, Dose-reduced Open Label) (Experimental): Following participation in the Double-blind Treatment Period, if an intolerable AE occurred, LINZESS® 72 μg capsules, orally, once daily up to Week 52 for participants with CIC.
  Interventions: Drug: Linaclotide
- LINZESS® 72 μg (IBS-C, Dose-reduced Open Label) (Experimental): Following participation in the Double-blind Treatment Period, if an intolerable AE occurred, LINZESS® 72 μg capsules, orally, once daily up to Week 52 for participants with IBS-C.
  Interventions: Drug: Linaclotide

INTERVENTIONS:
Drug: Linaclotide — Linaclotide capsules, orally, once daily.
  Other Names: LINZESS®

SUMMARY:
The primary objective of this study is to assess the potential of LINZESS® (linaclotide) treatment to induce the development of anti-drug antibodies (ADAs). The secondary objectives are to provide additional evidence supporting the long-term safety and efficacy of linaclotide in adult irritable bowel syndrome with constipation (IBS-C) and chronic idiopathic constipation (CIC) participants and to evaluate lower doses of linaclotide.

DETAILED DESCRIPTION:
This study includes up to a 3-week Screening Period, followed by a 52-week treatment period. Participants with CIC meeting the entry criteria received linaclotide 145 μg capsules, orally, once daily and participants with IBS-C meeting the entry criteria received linaclotide 290 μg capsules, orally, once daily. Participants with intolerable Adverse Events (AEs), following resolution of the AEs, could be randomized to receive 290 μg, 145 μg, or the lower dose of 72 μg linaclotide oral capsules for IBS-C; and 145 μg or 72 μg for CIC. Participants who experienced further intolerable AEs after the randomization could be transitioned to open-label 72 μg linaclotide.

ELIGIBILITY:
Inclusion Criteria:

* Participants meet the Rome III criteria for IBS-C or CIC:
* IBS-C Criteria: the participant must meet the following 2 criteria (A and B).

A. IBS Criteria: The participant must have abdominal pain or discomfort at least 3 days per month in the 3 months before diagnosis (with symptom onset at least 6 months before diagnosis) associated with 2 or more of the following:

1. Improvement with defecation.
2. Onset associated with a change in frequency of stool.
3. Onset associated with a change in form (appearance) of stool. B. Stool Consistency Requirement: During the 3 months before diagnosis in the absence of laxative or enema use, the patient has hard or lumpy stools (Bristol Stool Form Scale [BSFS] score 1 or 2) with at least 25% of bowel movements (BMs) and has loose or mushy stools (BSFS 5 or 6) with <25% of BMs.

   * CIC Criteria: the participant must meet the following 3 criteria (A, B, and C):

A. Participant meets 2 or more of the following criteria for 3 months before the diagnosis with symptom onset at least 6 months before diagnosis:

1. Straining during at least 25% of defecations.
2. Lumpy or hard stools in at least 25% of defecations.
3. Sensation of incomplete evacuation for at least 25% of defecations.
4. Sensation of anorectal obstruction/blockage for at least 25% of defecations.
5. Manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor).
6. Fewer than 3 defecations per week. B. Loose stools are rarely present without the use of laxatives. C. Insufficient criteria for irritable bowel syndrome. (The criteria for IBS are provided in Point A under IBS Criteria, above).

   * Participant meets the colonoscopy requirements, which are modified from the Summary of the US-Multi-Society Task Force on Colorectal Cancer and other Colonoscopy Requirements.
   * Participant has successfully completed protocol procedures (with no clinically significant findings).

Exclusion Criteria:

* At Day 1 visit, the participant reports having 6 or more spontaneous bowel movements (SBMs) in the week prior to screening.
* At Day 1 visit, the participant reports having any SBMs that were watery (BSFS=7) or more than 1 SBM that was mushy (BSFS=6) in the week prior to screening.
* Participant has a structural abnormality of the gastrointestinal (GI) tract or a disease or condition that can affect GI motility.
* Participant has any protocol excluded or clinically significant medical or surgical history that would limit the patient's ability to complete or participate in this clinical trial or could confound the study assessments.
* Participant has ever received linaclotide as a treatment (including commercially-available product) or has been randomized into any clinical study in which linaclotide was a treatment. (participant who enrolled into linaclotide clinical studies conducted prior or during this study but failed to be randomized are eligible for the current study).
* Participant has ever received plecanatide, SP-333, or has participated in a plecanatide clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wieslaw Bochenek, Study Director — Allergan
Locations (78):
- United States (78):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - North Alabama Research Center, LLC, Athens, Alabama
  - Alliance Clinical Research, Childersburg, Alabama
  - G & L Research, LLC, Foley, Alabama
  - Radiant Research, Inc., Chandler, Arizona
  - Radiant Research, Inc., Scottsdale, Arizona
  - Clinical Research Institute of Arizona, LLC, Surprise, Arizona
  - Clinical Research Consortium, Tempe, Arizona
  - Desert Sun Clinical Research, LLC., Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Global Clinical Trials LLC, Costa Mesa, California
  - Diagnamics Inc, Encinitas, California
  - MD Studies, Inc., Fountain Valley, California
  - Research Center of Fresno, Inc., Fresno, California
  - VVCRD Clinical Research, Garden Grove, California
  - Facey Medical Foundation, Mission Hills, California
  - Clinical Trials Research, Sacramento, California
  - Northern California Research, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Precision Research Institute, San Diego, California
  - Empire Clinical Research, Upland, California
  - Lynn Institute of Denver, Denver, Colorado
  - ZASA Clinical Research, Boynton Beach, Florida
  - Meridien Research, Bradenton, Florida
  - Clinical Research of Brandon LLC, Brandon, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Eastern Research, Inc., Hialeah, Florida
  - Center for Advanced Gastroenterology, Maitland, Florida
  - Florida Medical Center and Research, Inc., Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Accord Clinical Research, Port Orange, Florida
  - Meridien Research, St. Petersburg, Florida
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Northwest Clinical Trials, Boise, Idaho
  - Rockford Gastroenterology Associates, Rockford, Illinois
  - Iowa Digestive Center, PC, Clive, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Heartland Research Associates, LLC, Newton, Kansas
  - Health Science Research Center, Pratt, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - KAMP Medical Research Inc, Natchitoches, Louisiana
  - Coastal Research Associates, Inc., South Weymouth, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Aa Mrc Llc, Flint, Michigan
  - Beyer Research, Kalamazoo, Michigan
  - The Center for Clinical Trials, Inc., Biloxi, Mississippi
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Digestive Health Associates, Reno, Nevada
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Manhattan Medical Research Practice PLLC, New York, New York
  - DiGiovanna Institute for Medical Education & Research, North Massapequa, New York
  - UNC Health Care, University of North Carolina Medical Center, Memorial Hospital, Chapel Hill, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Northstate Clinical Research, Lenoir, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Clinical Inquest Center LTD, Dayton, Ohio
  - Dayton Gastroenterology, Inc., Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, INC, Pittsburgh, Pennsylvania
  - Montgomery Medical, Inc., Smithfield, Pennsylvania
  - Partners In Clinical Research, Cumberland, Rhode Island
  - Greenville Pharmaceutical Research, Inc., Greenville, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Houston Endoscopy & Research Center, Houston, Texas
  - Research Across America, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 828 participants were enrolled, 2 participants were enrolled but did not receive study treatment and were not included in any analysis populations.
Pre-assignment Details: 826 participants received LINZESS® 145μg [CIC] and 290μg [IBS-C] in the Open Label Treatment Period. Out of 826, 114 participants were randomized in the Double-blind Treatment Period and 57 out of 114 participants received 72 μg in the Dose-reduced Open Label Treatment Period due to intolerable AEs.
Groups:
- LINZESS® 145 μg (CIC, Open Label): LINZESS® 145 μg capsules, orally, once daily for up to 52 weeks for participants with chronic idiopathic constipation (CIC). If an intolerable adverse event (AE) occurred participants could be randomized to the Double-blind Treatment Period.
- LINZESS® 290 μg (IBS-C, Open Label): LINZESS® 290 μg capsules, orally, once daily for up to 52 weeks for participants with irritable bowel syndrome with constipation (IBS-C). If an intolerable AE occurred participants could be randomized to the Double-blind Treatment Period.
Period: Open-label Treatment Period
Arm/Group | LINZESS® 145 μg (CIC, Open Label) | LINZESS® 290 μg (IBS-C, Open Label) | LINZESS® 290 μg (IBS-C, Double Blind) | LINZESS® 145 μg (IBS-C, Double Blind) | LINZESS® 72 μg (IBS-C, Double Blind) | LINZESS® 145 μg (CIC, Double Blind) | LINZESS® 72 μg (CIC, Double Blind) | LINZESS® 72 μg (CIC, Dose-reduced Open Label) | LINZESS® 72 μg (IBS-C, Dose-reduced Open Label)
Started | 508 | 318 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed (Out of 384 participants who discontinued, 114 continued to Double-blind Treatment Period.) | 276 (Participants were not randomized to Double-blind Treatment Period.) | 166 (Participants were not randomized to Double-blind Treatment Period.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 232 | 152 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 97 | 79 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 14 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 43 | 28 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 51 | 29 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 10 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 7 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Miscellaneous Reasons | 10 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Double-blind Treatment Period
Arm/Group | LINZESS® 145 μg (CIC, Open Label) | LINZESS® 290 μg (IBS-C, Open Label) | LINZESS® 290 μg (IBS-C, Double Blind) | LINZESS® 145 μg (IBS-C, Double Blind) | LINZESS® 72 μg (IBS-C, Double Blind) | LINZESS® 145 μg (CIC, Double Blind) | LINZESS® 72 μg (CIC, Double Blind) | LINZESS® 72 μg (CIC, Dose-reduced Open Label) | LINZESS® 72 μg (IBS-C, Dose-reduced Open Label)
Started | 0 | 0 | 18 | 18 | 16 | 32 | 30 | 0 | 0
Completed (Out of 88 participants who discontinued, 57 continued to Dose-reduced Open Label Treatment Period.) | 0 | 0 | 1 (Participants did not enter Dose-reduced Open Label Treatment Period.) | 3 (Participants did not enter Dose-reduced Open Label Treatment Period.) | 7 (Participants did not enter Dose-reduced Open Label Treatment Period.) | 6 (Participants did not enter Dose-reduced Open Label Treatment Period.) | 9 (Participants did not enter Dose-reduced Open Label Treatment Period.) | 0 | 0
Not Completed | 0 | 0 | 17 | 15 | 9 | 26 | 21 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 14 | 12 | 6 | 22 | 20 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 0 | 0 | 1 | 3 | 3 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Non-compliance with Study Drug | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Dose-reduced Open Label Treatment Period
Arm/Group | LINZESS® 145 μg (CIC, Open Label) | LINZESS® 290 μg (IBS-C, Open Label) | LINZESS® 290 μg (IBS-C, Double Blind) | LINZESS® 145 μg (IBS-C, Double Blind) | LINZESS® 72 μg (IBS-C, Double Blind) | LINZESS® 145 μg (CIC, Double Blind) | LINZESS® 72 μg (CIC, Double Blind) | LINZESS® 72 μg (CIC, Dose-reduced Open Label) | LINZESS® 72 μg (IBS-C, Dose-reduced Open Label)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 26
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 15
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Non-compliance with Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other Miscellaneous Reasons | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants in the screened population (all participants who had signed an informed consent form (ICF) for the study and received a patient identification number) who received ≥ 1 administration of study treatment.
Groups:
- LINZESS® 145 μg (CIC, Open Label): LINZESS® 145 μg capsules, orally, once daily for up to 52 weeks for participants with CIC. If an intolerable AE occurred participants could be randomized to the Double-blind Treatment Period.
- Total: Total of all reporting groups
Arm/Group | LINZESS® 145 μg (CIC, Open Label) | LINZESS® 290 μg (IBS-C, Open Label) | Total
Number analyzed (Participants) | 508 | 318 | 826
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (15.3) | 45.2 (13.9) | 47.9 (14.9)
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 140 | 120 | 260
  >=40 to <65 years | 274 | 170 | 444
  >=65 years | 94 | 28 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 410 | 259 | 669
  Male | 98 | 59 | 157
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 348 | 227 | 575
  Black or African American | 135 | 68 | 203
  Asian | 19 | 17 | 36
  American Indian or Alaska Native | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Multiple Races | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 124 | 76 | 200
  Not Hispanic or Latino | 384 | 242 | 626

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Treatment-Related Anti-Drug Antibodies (ADA) in Serum
Description: Participants who met either of the following criteria: 1) treatment-induced ADA-positive (≥ 1 postbaseline ADA-positive sample) for baseline ADA negative or ADA-undetermined participants or 2) treatment-boosted ADA-positive (≥ 1 postbaseline ADA-positive sample with titer values ≥ 4-fold the baseline titer value) for baseline ADA-positive participants were reported as a ADA positive responder.
Time Frame: Baseline (Day 1) up to 52 weeks or 8 months post last dose if ADA positive at Week 52 (approximately 84 weeks)
Population: Safety population included all participants in the screened population (all participants who had signed an informed consent form (ICF) for the study and received a patient identification number) who received ≥ 1 administration of study treatment. Participants with ≥ 1 assessable postbaseline sample were analyzed (ADA-undetermined excluded).
Measure: Count of Participants; unit: Participants
Arm/Group | LINZESS® 145 μg (CIC, Open Label) | LINZESS® 290 μg (IBS-C, Open Label)
Number analyzed (Participants) | 498 | 309
Participants | 3 | 1

2. Secondary Outcome: Change From Baseline in Participant's Assessment of Constipation Severity
Description: Participants rated constipation severity during the previous 7 days on a 5-point ordinal scale where, 1=None, 2=Mild, 3=Moderate, 4=Severe and 5=Very Severe. Higher scores indicate greater severity. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Weeks 2, 4, 12, 26, 40 and 52 (Open Label Treatment Period)
Population: Intent to Treat (ITT) population included all participants in the safety population who had ≥ 1 postbaseline assessment for any efficacy or health outcomes parameter. Number analyzed were the participants with analysis values at both baseline and postbaseline during the specified time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LINZESS® 145 μg (CIC, Open Label) | LINZESS® 290 μg (IBS-C, Open Label)
Number analyzed (Participants) | 503 | 311
score on a scale
  Baseline | 3.5 (0.8) | 3.4 (0.8)
  Change from Baseline at Week 2: number analyzed (Participants) | 496 | 307
  Change from Baseline at Week 2 | -1.1 (1.1) | -1.2 (1.1)
  Change from Baseline at Week 4: number analyzed (Participants) | 476 | 299
  Change from Baseline at Week 4 | -1.3 (1.1) | -1.3 (1.1)
  Change from Baseline at Week 12: number analyzed (Participants) | 434 | 265
  Change from Baseline at Week 12 | -1.4 (1.1) | -1.3 (1.2)
  Change from Baseline at Week 26: number analyzed (Participants) | 360 | 230
  Change from Baseline at Week 26 | -1.4 (1.1) | -1.3 (1.1)
  Change from Baseline at Week 40: number analyzed (Participants) | 318 | 198
  Change from Baseline at Week 40 | -1.6 (1.1) | -1.3 (1.0)
  Change from Baseline at Week 52: number analyzed (Participants) | 301 | 183
  Change from Baseline at Week 52 | -1.6 (1.1) | -1.5 (1.1)

3. Secondary Outcome: Change From Baseline in Participant Assessment of Irritable Bowel Syndrome (IBS) Symptom Severity for Participants With Irritable Bowel Syndrome With Constipation (IBS-C)
Description: Participants rated IBS symptoms severity during the previous 7 days on a 5-point ordinal scale where, 1=None, 2=Mild, 3=Moderate, 4=Severe and 5=Very severe. Higher scores indicate greater severity. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 2, 4, 12, 26, 40 and 52 (Open Label Treatment Period)
Population: ITT population consisted of all participants in the safety population who had ≥ 1 postbaseline assessment for any efficacy or health outcomes parameter. Number analyzed were the participants with analysis values at both baseline and postbaseline during the specified time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LINZESS® 290 μg (IBS-C, Open Label)
Number analyzed (Participants) | 311
score on a scale
  Baseline: number analyzed (Participants) | 309
  Baseline | 3.4 (0.7)
  Change from Baseline at Week 2: number analyzed (Participants) | 305
  Change from Baseline at Week 2 | -1.0 (1.1)
  Change from Baseline at Week 4: number analyzed (Participants) | 298
  Change from Baseline at Week 4 | -1.1 (1.0)
  Change from Baseline at Week 12: number analyzed (Participants) | 264
  Change from Baseline at Week 12 | -1.2 (1.1)
  Change from Baseline at Week 26: number analyzed (Participants) | 230
  Change from Baseline at Week 26 | -1.2 (1.0)
  Change from Baseline at Week 40: number analyzed (Participants) | 198
  Change from Baseline at Week 40 | -1.2 (1.0)
  Change from Baseline at Week 52: number analyzed (Participants) | 184
  Change from Baseline at Week 52 | -1.3 (1.0)

4. Secondary Outcome: Change From Baseline in Degree of Relief of IBS Symptoms for Participants With IBS-C
Description: Participants rated degree of relief of IBS symptoms during previous 7 days on a 7-point balanced ordinal scale where, 1=completely relieved, 2=considerably relieved, 3=somewhat relieved, 4=unchanged, 5=somewhat worse, 6=considerably worse and 7=as bad as I can imagine. Lower scores indicate greater relief. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Weeks 2, 4, 12, 26, 40 and 52 (Open Label Treatment Period)
Population: Intent-to-treat (ITT) population included all participants in the safety population who had ≥ 1 postbaseline assessment for any efficacy or health outcomes parameter. Number analyzed were the participants with analysis values at both baseline and postbaseline during the specified time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LINZESS® 290 μg (IBS-C, Open Label)
Number analyzed (Participants) | 311
score on a scale
  Baseline: number analyzed (Participants) | 308
  Baseline | 4.2 (0.8)
  Change from Baseline at Week 2: number analyzed (Participants) | 304
  Change from Baseline at Week 2 | -1.4 (1.3)
  Change from Baseline at Week 4: number analyzed (Participants) | 297
  Change from Baseline at Week 4 | -1.6 (1.3)
  Change from Baseline at Week 12: number analyzed (Participants) | 263
  Change from Baseline at Week 12 | -1.8 (1.3)
  Change from Baseline at Week 26: number analyzed (Participants) | 229
  Change from Baseline at Week 26 | -1.8 (1.3)
  Change from Baseline at Week 40: number analyzed (Participants) | 197
  Change from Baseline at Week 40 | -1.9 (1.3)
  Change from Baseline at Week 52: number analyzed (Participants) | 183
  Change from Baseline at Week 52 | -1.8 (1.3)

5. Secondary Outcome: IBS Treatment Satisfaction Assessment Postbaseline for Participants With IBS-C
Description: Participants rated degree of satisfaction with the LINZESS®'s ability to relieve IBS symptoms on a 5-point ordinal scale where, 1=Not at all satisfied, 2=A little satisfied, 3=Moderately satisfied, 4=Quite satisfied and 5=Very satisfied. Higher scores indicate greater satisfaction.
Time Frame: Weeks 2, 4, 12, 26, 40 and 52 (Open Label Treatment Period)
Population: ITT population included all participants in the safety population who had ≥ 1 postbaseline assessment for any efficacy or health outcomes parameter. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LINZESS® 290 μg (IBS-C, Open Label)
Number analyzed (Participants) | 311
score on a scale
  Week 2: number analyzed (Participants) | 306
  Week 2 | 3.3 (1.2)
  Week 4: number analyzed (Participants) | 299
  Week 4 | 3.6 (1.1)
  Week 12: number analyzed (Participants) | 265
  Week 12 | 3.7 (1.1)
  Week 26: number analyzed (Participants) | 230
  Week 26 | 3.7 (1.1)
  Week 40: number analyzed (Participants) | 198
  Week 40 | 3.7 (1.1)
  Week 52: number analyzed (Participants) | 184
  Week 52 | 3.8 (1.1)

6. Secondary Outcome: Constipation Treatment Satisfaction Assessment Postbaseline for Participants With Chronic Idiopathic Constipation (CIC)
Description: Participants rated degree of satisfaction with LINZESS®'s ability to relieve constipation symptoms on a 5-point ordinal scale where 1=Not at all satisfied, 2=A little satisfied, 3=Moderately satisfied, 4=Quite satisfied and 5=Very satisfied. Higher scores indicate greater satisfaction.
Time Frame: Weeks 2, 4, 12, 26, 40 and 52 (Open Label Treatment Period)
Population: ITT population consisted of all participants in the safety population who had ≥ 1 postbaseline assessment for any efficacy or health outcomes parameter. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LINZESS® 145 μg (CIC, Open Label)
Number analyzed (Participants) | 503
score on a scale
  Week 2: number analyzed (Participants) | 495
  Week 2 | 3.4 (1.2)
  Week 4: number analyzed (Participants) | 476
  Week 4 | 3.5 (1.2)
  Week 12: number analyzed (Participants) | 435
  Week 12 | 3.7 (1.1)
  Week 26: number analyzed (Participants) | 359
  Week 26 | 3.8 (1.1)
  Week 40: number analyzed (Participants) | 318
  Week 40 | 3.9 (1.1)
  Week 52: number analyzed (Participants) | 301
  Week 52 | 4.0 (1.1)

7. Secondary Outcome: Number of Participants With Recurrence of Diarrhea
Description: Participant reporting any instance of diarrhea during the Double-blind Treatment Period.
Time Frame: From first dose in the Double-blind Treatment Period to Week 52
Population: Double-blind safety population consisted of all participants in the randomized population who received ≥ 1 dose of study treatment during the Double-blind Treatment Period. Number of Participants Analyzed were the participants reporting intolerable diarrhea during the Open-label Treatment Period.
Measure: Count of Participants; unit: Participants
Arm/Group | LINZESS® 290 μg (IBS-C, Double Blind) | LINZESS® 145 μg (IBS-C, Double Blind) | LINZESS® 72 μg (IBS-C, Double Blind) | LINZESS® 145 μg (CIC, Double Blind) | LINZESS® 72 μg (CIC, Double Blind)
Number analyzed (Participants) | 17 | 17 | 16 | 29 | 29
Participants | 11 | 12 | 5 | 19 | 18
Statistical Analysis 1: Comparison: LINZESS® 290 μg (IBS-C, Double Blind) vs LINZESS® 145 μg (IBS-C, Double Blind); LINZESS® 145 μg versus (vs) LINZESS® 290 μg; Test type: Superiority; p = 1.0000, Fisher's Exact Test; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.3 to 5.5]
Statistical Analysis 2: Comparison: LINZESS® 290 μg (IBS-C, Double Blind) vs LINZESS® 72 μg (IBS-C, Double Blind); LINZESS® 72 μg vs LINZESS® 290 μg; Test type: Superiority; p = 0.0844, Fisher's Exact Test; Odds Ratio (OR) = 0.2, 95% CI 2-sided [0.1 to 1.1]
Statistical Analysis 3: Comparison: LINZESS® 145 μg (CIC, Double Blind) vs LINZESS® 72 μg (CIC, Double Blind); LINZESS® 72 μg vs LINZESS® 145 μg; Test type: Superiority; p = 1.0000, Fisher's Exact Test; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.3 to 2.5]

8. Secondary Outcome: Number of Participants With Recurrence of Intolerable Diarrhea
Description: Participants reporting any instance of intolerable diarrhea during the Double-blind Treatment Period (Non-responder otherwise). Only includes participants reporting intolerable diarrhea during the Open-label Treatment Period.
Time Frame: From first dose in the Double-blind Treatment Period to Week 52
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | LINZESS® 290 μg (IBS-C, Double Blind) | LINZESS® 145 μg (IBS-C, Double Blind) | LINZESS® 72 μg (IBS-C, Double Blind) | LINZESS® 145 μg (CIC, Double Blind) | LINZESS® 72 μg (CIC, Double Blind)
Number analyzed (Participants) | 17 | 17 | 16 | 29 | 29
Participants | 10 | 11 | 4 | 19 | 17
Statistical Analysis 1: Comparison: LINZESS® 290 μg (IBS-C, Double Blind) vs LINZESS® 145 μg (IBS-C, Double Blind); LINZESS® 145 μg vs LINZESS® 290 μg; Test type: Superiority; p = 1.0000, Fisher's Exact Test; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.3 to 5.1]
Statistical Analysis 2: Comparison: LINZESS® 290 μg (IBS-C, Double Blind) vs LINZESS® 72 μg (IBS-C, Double Blind); LINZESS® 72 μg vs LINZESS® 290 μg; Test type: Superiority; p = 0.0799, Fisher's Exact Test; Odds Ratio (OR) = 0.2, 95% CI 2-sided [0.1 to 1.0]
Statistical Analysis 3: Comparison: LINZESS® 145 μg (CIC, Double Blind) vs LINZESS® 72 μg (CIC, Double Blind); LINZESS® 72 μg vs LINZESS® 145 μg; Test type: Superiority; p = 0.7871, Fisher's Exact Test; Odds Ratio (OR) = 0.7, 95% CI 2-sided [0.3 to 2.2]

9. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAE)
Description: An adverse event is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is an AE that occurred after receiving the first dose of investigational product or an AE present prior to first dose but increased in severity during the Treatment Period.
Time Frame: From first dose of study treatment up to Week 52
Population: Safety population included all participants in the screened population who received ≥ 1 administration of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | LINZESS® 145 μg (CIC, Open Label) | LINZESS® 290 μg (IBS-C, Open Label)
Number analyzed (Participants) | 508 | 318
percentage of participants | 62.6 | 66.0

10. Secondary Outcome: Time to First Recurrence of Diarrhea
Description: Time to first recurrence of diarrhea was defined as event/censored date - double-blind start date + 1, where event date (responders) = first recurrence of diarrhea date during the double-blind treatment period; censoring date (non-responders) = double-blind end date. Only includes participants reporting intolerable diarrhea during the open-label treatment period.
Time Frame: From first dose in the Double-blind Treatment Period to Week 52
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | LINZESS® 290 μg (IBS-C, Double Blind) | LINZESS® 145 μg (IBS-C, Double Blind) | LINZESS® 72 μg (IBS-C, Double Blind) | LINZESS® 145 μg (CIC, Double Blind) | LINZESS® 72 μg (CIC, Double Blind)
Number analyzed (Participants) | 17 | 17 | 16 | 29 | 29
days | 19.0 [2.0 to 64.0] | 15.0 [2.0 to 96.0] | NA [21.0 to NA] — Median and upper limit of CI was not reached due to low number of participants with events. | 4.0 [1.0 to NA] — Upper limit of CI was not reached due to low number of participants with events. | 9.0 [3.0 to NA] — Upper limit of CI was not reached due to low number of participants with events.
Statistical Analysis 1: Comparison: LINZESS® 290 μg (IBS-C, Double Blind) vs LINZESS® 145 μg (IBS-C, Double Blind); LINZESS® 145 μg vs LINZESS® 290 μg; Test type: Superiority; p = 0.9930, Log-Rank Test; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.42 to 2.19]
Statistical Analysis 2: Comparison: LINZESS® 290 μg (IBS-C, Double Blind) vs LINZESS® 72 μg (IBS-C, Double Blind); LINZESS® 72 μg vs LINZESS® 290 μg; Test type: Superiority; p = 0.0247, Log-Rank Test; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.11 to 0.89]
Statistical Analysis 3: Comparison: LINZESS® 145 μg (CIC, Double Blind) vs LINZESS® 72 μg (CIC, Double Blind); LINZESS® 72 μg vs LINZESS® 145 μg; Test type: Superiority; p = 0.5149, Log-Rank Test; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.41 to 1.50]

11. Secondary Outcome: Time to First Recurrence of Intolerable Diarrhea
Description: Time to first recurrence of intolerable diarrhea was defined as event/censored date - double-blind start date + 1, where event date (responders) = first recurrence of intolerable diarrhea date during the double-blind treatment period; censoring date (non-responders) = double-blind end date. Only includes participants reporting intolerable diarrhea during the open-label treatment period.
Time Frame: From first dose in the Double-blind Treatment Period to Week 52
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | LINZESS® 290 μg (IBS-C, Double Blind) | LINZESS® 145 μg (IBS-C, Double Blind) | LINZESS® 72 μg (IBS-C, Double Blind) | LINZESS® 145 μg (CIC, Double Blind) | LINZESS® 72 μg (CIC, Double Blind)
Number analyzed (Participants) | 17 | 17 | 16 | 29 | 29
days | 19.0 [2.0 to NA] — Upper limit of CI was not reached due to low number of participants with events. | 18.0 [2.0 to NA] — Upper limit of CI was not reached due to low number of participants with events. | NA [55.0 to NA] — Median and upper limit of CI was not reached due to low number of participants with events. | 8.0 [1.0 to 254.0] | 9.0 [3.0 to NA] — Upper limit of CI was not reached due to low number of participants with events.
Statistical Analysis 1: Comparison: LINZESS® 290 μg (IBS-C, Double Blind) vs LINZESS® 145 μg (IBS-C, Double Blind); LINZESS® 145 μg vs LINZESS® 290 μg; Test type: Superiority; p = 0.9519, Log-Rank Test; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.39 to 2.18]
Statistical Analysis 2: Comparison: LINZESS® 290 μg (IBS-C, Double Blind) vs LINZESS® 72 μg (IBS-C, Double Blind); LINZESS® 72 μg vs LINZESS® 290 μg; Test type: Superiority; p = 0.0234, Log-Rank Test; Hazard Ratio (HR) = 0.27, 95% CI 2-sided [0.08 to 0.87]
Statistical Analysis 3: Comparison: LINZESS® 145 μg (CIC, Double Blind) vs LINZESS® 72 μg (CIC, Double Blind); LINZESS® 72 μg vs LINZESS® 145 μg; Test type: Superiority; p = 0.4518, Log-Rank Test; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.39 to 1.47]

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to 1 day post last dose for non-serious adverse events and up to 30 days post last dose of study treatment for serious adverse events (Up to 56 Weeks)
Description: Adverse Events were monitored/assessed according to indication (CIC and IBS-C), irrespective of the dose level, and cannot be reported for each dose separately.
Groups:
- LINZESS® 145 μg (CIC): LINZESS® 145 μg capsules, orally, once daily for up to 52 weeks for participants with CIC. If an Intolerable AE occurred participants could be randomized to the Double-blind Treatment Period (145 μg or 72 μg) or entered the Dose-reduced 72 μg Open Label Period.
- LINZESS® 290 μg (IBS-C): LINZESS® 290 μg capsules, orally, once daily for up to 52 weeks for participants with IBS-C. If an intolerable AE occurred participants could be randomized to the Double-blind Treatment Period (290 μg, 145 μg or 72 μg) or entered the Dose-reduced 72 μg Open Label Period.
Arm/Group | LINZESS® 145 μg (CIC) | LINZESS® 290 μg (IBS-C)
All-Cause Mortality (participants affected / at risk) | 1/508 | 0/318
Serious Adverse Events (participants affected / at risk) | 16/508 | 6/318
Other Adverse Events (participants affected / at risk) | 133/508 | 122/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LINZESS® 145 μg (CIC) (N=508) | LINZESS® 290 μg (IBS-C) (N=318)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 2 | 0
Thyroid mass (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Allergy to venom (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibrin D dimer increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Hemiplegic migraine (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LINZESS® 145 μg (CIC) (N=508) | LINZESS® 290 μg (IBS-C) (N=318)
Diarrhoea (Gastrointestinal disorders) | 130 | 116
Flatulence (Gastrointestinal disorders) | 11 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT02590432/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT02590432/SAP_001.pdf